CLINICAL TRIAL: NCT06396208
Title: "Quick-starting" of a Quadriphasic Contraceptive Pills, 1 - 3 mg Estradiol Valerate/ 2 - 3 mg Dienogest VS 20 mcg Ethinylestradiol/75 mcg Gestodene Focusing on Ovulation Inhibition: A Single-blind, Randomized Controlled, Non-inferiority Trial
Brief Title: "Quick-starting" of a Quadriphasic Contraceptive Pills, 1 - 3 mg Estradiol Valerate/ 2 - 3 mg Dienogest VS 20 mcg Ethinylestradiol/75 mcg Gestodene Focusing on Ovulation Inhibition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB0838/66
Record Dates: First submitted 2024-04-25; First posted 2024-05-02 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-04

CONDITIONS: Ultrasound Finding: Ovulation Inhibition, Ovarian Activities; Cervical Mucus; Serum Hormonal Profile
Keywords: Quick starting contraception; Quadriphasic combined hormonal contraceptive pill(s); Estradiol valerate/Dienogest; Ovulation inhibition
MeSH Terms: interventions — dienogest; Ethinyl Estradiol; Gestodene

STUDY DESIGN:
Intervention Model Description: Ethinylestradiol (EE) 20 mcg/Gestodene 75 mcg (21/7) as control group Quadriphasic Estradiol valerate 1 - 3 mg/ Dienogest 2 - 3 mg (26/2) as intervention group
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadriphasic Estradiol valerate 1 - 3 mg/ Dienogest 2 - 3 mg (26/2) (Experimental): Completing a pack (28 pills) of Quadriphasic Estradiol valerate 1 - 3 mg/ Dienogest 2 - 3 mg (26/2), starting on day 7-9 of menstrual cycle
  Interventions: Drug: Quadriphasic Estradiol valerate 1 - 3 mg/ Dienogest 2 - 3 mg (26/2)
- Ethinylestradiol (EE) 20 mcg/Gestodene 75 mcg (21/7) (Active Comparator): Completing a pack (28 pills) of Ethinylestradiol (EE) 20 mcg/Gestodene 75 mcg (21/7), starting on day 7-9 of menstrual cycle
  Interventions: Drug: Ethinylestradiol (EE) 20 mcg/Gestodene 75 mcg (21/7)

INTERVENTIONS:
Drug: Quadriphasic Estradiol valerate 1 - 3 mg/ Dienogest 2 - 3 mg (26/2) — Completing a pack (28 pills) of Quadriphasic Estradiol valerate 1 - 3 mg/ Dienogest 2 - 3 mg (26/2), starting on day 7-9 of menstrual cycle
  Arms: Quadriphasic Estradiol valerate 1 - 3 mg/ Dienogest 2 - 3 mg (26/2)
Drug: Ethinylestradiol (EE) 20 mcg/Gestodene 75 mcg (21/7) — Completing a pack (28 pills) of Ethinylestradiol (EE) 20 mcg/Gestodene 75 mcg (21/7), starting on day 7-9 of menstrual cycle
  Arms: Ethinylestradiol (EE) 20 mcg/Gestodene 75 mcg (21/7)

SUMMARY:
The goal of this clinical trial is to learn if Estetrol/Drospirenone inhibit ovulation in quick-starting method. It will also learn about the safety of Estetrol/Drospirenone. The main questions it aims to answer are:

Does Estradiol valerate/Dienogest inhibit ovulation inferior to Ethinyl estradiol/Gestodene when starting on Day 7-9 of menstrual cycle? What are the impacts of Estradiol valerate/Dienogest on ovarian activities when starting on Day 7-9 of menstrual cycle? How does the cervical mucus change when starting Estradiol valerate/Dienogest on Day 7-9 of menstrual cycle? What are the adverse effects when starting Estradiol valerate/Dienogest on Day 7-9 of menstrual cycle? Researchers will compare Estradiol valerate/Dienogest to Ethinyl estradiol/Gestodene to see if Estradiol valerate/Dienogest inhibit ovulation in quick-starting method.

DETAILED DESCRIPTION:
Take Estradiol valerate/Dienogest or Ethinyl estradiol/Gestodene starting on day 7-9 of menstrual cycle then every day for 1 pack of the pills.

Visit the clinic on day 1-2, day 7-9, and then every 2-7 days according to ultrasound finding (ovarian activities) until completing of pills to investigate

* Transvaginal ultrasound
* Cervical mucus
* Serum hormonal profiles.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 - 45 years old
* Body mass index 18-30 kg/m²
* Menstrual interval within 24 - 38 days
* Absence of history of estrogen or progestin allergy and Absence of these compatibles with U.S. medical eligibility criteria category 3 - 4
* Consent to use condom as contraception or have been sterilized

Exclusion Criteria:

* History of estrogen, progestin or testosterone use within 3 months
* Current pregnant or within 3 months of breastfeeding
* Having ovarian cyst(s) or tumor(s)
* Being a cervical cancer patient or having precancerous cervical lesion

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Rate of ovulation inhibition and classify ovarian activities using transvaginal ultrasound | 34-36 days
  Visit the clinic on day 1-2, day 7-9, and then every 2-7 days according to ultrasound finding until completing a package of pills
  * Ultrasound will be perform by the researcher (Dr. Sirarat Itthipuripat) using transvaginal probe to all volunteers.
  * To monitor a leading ovarian follicle or follicle-like structures (FLS), that the ultrasound characteristic is the largest hypoechoic part (follicle) among both ovaries, to classify the ovarian activity by modified Hoogland's score (combined the result with hormonal profile: Estradiol, Progesterone) and assess rate of ovulation, that identify from postovulatory image defined as follows:
  * Image observed after abrupt disappearance of FLS or
  * Image observed after reduction in size of the leading follicle > 4 mm at 2 consecutive visits or
  * Hemorrhagic or cystic corpus luteum
  * The detail in measuring the size of an FLS is the average of 3 longest sides perpendicular to each other in millimeter

SECONDARY OUTCOMES:
Level of serum hormonal profiles: Estradiol, Progesterone, LH | 34-36 days
  Visit the clinic on day 1-2, day 7-9, and then every 2-7 days according to ultrasound finding
  * Blood test to measure estrogen level in picogram/milliliter, progesterone level in nanogram/milliliter and LH level in International unit per liter
  * Volunteers will be placed in a 5 ml clot activator tube and sent to the endocrinology laboratory medical operation center within 30 minutes after blood draw.
Cervical mucus classification | 34-36 days
  Visit the clinic on day 1-2, day 7-9, and then every 2-7 days according to ultrasound finding
  * Using Tuberculin syringe 1 mL to suck cervical mucus from the endocervical canal (1 cm deep from external cervical os)
  * Assess the results of cervical mucus collected immediately according to WHO 2010, consisting of volume (milliliter), viscosity, ferning appearance, Spinnbarkeit (centimeter), and cellularity (cell/high power field), under microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Somsook Santibenchakul, Master, Study Director — Obstetric and gynecology department, Faculty of medicine, Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No